CLINICAL TRIAL: NCT05992753
Title: Mothers' Breast Milk Expression Experiences, Infant Feeding Attitudes and Perceived Social Support Levels in the Early Postpartum Period: A Cross-sectional Study in Turkish Population
Brief Title: Mothers' Breast Milk Expression Experiences, Infant Feeding Attitudes and Perceived Social Support Levels
Status: Completed | Type: Observational
Sponsor: Halic University (Other)
Collaborators: Istanbul Arel University (Other); Istanbul University - Cerrahpasa (Other); Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2023-07-31; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Breastfeeding; Breast Milk Expression; Feeding Behavior; Support, Family
MeSH Terms: conditions — Breast Feeding; Breast Milk Expression; Feeding Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire application — The research data were collected from 455 mothers admitted to the postpartum and lactation unit of a city hospital in Istanbul between September and November 2022. The mothers to be included in the study sample were determined according to the non-probability sampling method, considering the inclusion criteria of the study. The research data were collected by the researchers face-to-face through a questionnaire that lasted about 10-20 minutes.

SUMMARY:
Background: Expressing breast milk in cases where breastfeeding is interrupted is important for infants to be fed breast milk however, many factors can affect mothers' breastfeeding experience, such as feeding attitudes and the level of social support. The aim of this study is to determine the relationship mothers' breast milk expression experience between infant feeding attitudes and perceived social support level.

Methods: This cross-sectional study was carried out in the postpartum and lactation unit of a city hospital in Istanbul, between September-November 2022. The study included 455 women who were volunteering to participate in the research, 18 years of age or older, in the 0-6 months postpartum period, having a living baby, continuing to breastfeed, and expressing breast milk at least once after birth. Data were collected with Mother-Baby Introductory Information Form, Breast Milk Expression Experience Measure (BMEE), Iowa Infant Feeding Attitude Scale (IIFAS), and Multidimensional Scale of Perceived Social Support (MSPSS). The data were analyzed using the SPSS-21 statistical software package.

The main questions it aims to answer are:

* Which characteristics affect mothers' breast milk expression experiences, infant feeding attitudes, and perceived social support levels in the early postpartum period?
* Is there a relationship between mothers' experiences of breast milk expression and their infant feeding attitudes and social support levels in the early postpartum period?

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research
* 18 years of age or older
* In the 0-6 month postpartum period
* Must have a living baby
* Must continue breastfeeding
* Must express breast milk at least once after birth

Exclusion Criteria:

* Feeding the infant formula only
* Having hearing and/or speech impairments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The research population consisted of women who were admitted to the postpartum and lactation units of a city hospital in Istanbul affiliated with the Turkish Ministry of Health. A power analysis was performed to determine the number of people to be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Mother-Baby Introductory Information Form | September 1st - November 30th 2022
  The form prepared by the researchers consists of 25 questions containing information about the mother, the infant, and the nutrition characteristics.
Breast Milk Expression Experience Measure (BMEE) | September 1st - November 30th 2022
  The BMEE, which was developed to determine the breast milk expression experience of mothers, consists of 11 items. The BMEE is a five-point Likert type, ranging from one (strongly disagree) to five (strongly agree). It has three sub-dimensions: social support, learning experience, and personal experience. When the mean of the total items' score is less than three, the breast milk expression experience of the mothers is evaluated as negative.
Iowa Infant Feeding Attitude Scale (IIFAS) | September 1st - November 30th 2022
  The scale was designed to evaluate women's attitudes towards breastfeeding and predict the duration of breastfeeding as well as the choice of infant feeding method. IIFAS consists of 17 items and is a five-point Likert type (one-strongly disagree to five-strongly agree). While nine items of the IIFAS contain positive attitudes about breastfeeding, the other eight items contain positive attitudes about formula feeding. The total IIFAS score can range from 17 to 85, with higher scores reflecting a positive attitude towards breastfeeding. Total IIFAS scores can be categorized into three groups: positive to breastfeeding (IIFAS score 70-85), neutral (IIFAS score 49-69), and positive to formula feeding (IIFAS score 17-48).
Multidimensional Scale of Perceived Social Support (MSPSS) | September 1st - November 30th 2022
  MSPSS subjectively assesses the adequacy of social support from three different sources (family, friends, and a significant other), consists of 12 items, and is a seven-point Likert type (one-very strongly disagree to seven-very strongly agree). The lowest score to be obtained from MSPSS is 12, and the highest score is 84. The higher the total score, the higher the perceived social support.

CONTACTS AND LOCATIONS:
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No